CLINICAL TRIAL: NCT02696928
Title: Feasibility of Methylene Blue-based Combination Therapy in the Radical Treatment of Adult Patients With Plasmodium Vivax Malaria in Ethiopia: a Randomised Controlled Pilot Trial
Brief Title: Methylene Blue Against Vivax Malaria in Ethiopia
Acronym: BlueAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of ethical approval in Ethiopia
Sponsor: Heidelberg University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Jimma University (Other)
Responsible Party: Principal Investigator, Olaf Mueller, Prof. Dr., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniHD007
Record Dates: First submitted 2016-02-02; First posted 2016-03-02 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — Combined Modality Therapy; 3,7-bis(diethylamino)phenothiazin-5-ium; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artemeter-Lumefantrine (combination therapy) (Other): 33 patients
  (standard of care)
  Interventions: Drug: Artemeter-Lumefantrine (combination therapy)
- Artemeter-Lumefantrine and Primaquine (combination therapy) (Active Comparator): 33 patients
  Interventions: Drug: Artemeter-Lumefantrine and Primaquine (combination therapy)
- Artemeter-Lumefantrine and MB (combination therapy) (Experimental): 33 patients
  Interventions: Drug: Artemeter-Lumefantrine and MB (combination therapy)

INTERVENTIONS:
Drug: Artemeter-Lumefantrine and MB (combination therapy) — AL first 3 days MB next 14 days
  Other Names: 3,7-bis(Dimethylamino)-phenothiazin-5-ium chloride; CID 6099
  Arms: Artemeter-Lumefantrine and MB (combination therapy)
Drug: Artemeter-Lumefantrine (combination therapy) — AL first 3 days
  Other Names: AL
  Arms: Artemeter-Lumefantrine (combination therapy)
Drug: Artemeter-Lumefantrine and Primaquine (combination therapy) — AL first 3 days PQ next 14 days
  Other Names: AL and PQ
  Arms: Artemeter-Lumefantrine and Primaquine (combination therapy)

SUMMARY:
Feasibility of methylene blue-based combination therapy in the radical treatment of adult patients with Plasmodium vivax malaria in Ethiopia: a randomised controlled pilot trial

Study rationale:

Elimination has become the goal of malaria programmes in an increasing number of endemic countries and regions. Primaquine (PQ) is the only registered drug for radical cure of Plasmodium vivax malaria. Prolonged PQ-based combination therapy carries safety concerns and resistance to chloroquine (CQ) and PQ is emerging. Methylene blue (MB) has recently been shown to be safe and effective in the treatment of Plasmodium falciparum malaria in West Africa. As there is evidence for MB probably being effective against the hypnozoites of Plasmodium vivax, MB-based drug regimens could be an alternative to PQ-based combination therapy in Plasmodium vivax malaria.

Study objectives:

The main objective of this trial is to study the feasibility of MB-based combination therapy in patients with uncomplicated P. vivax malaria in an endemic area of Ethiopia.

DETAILED DESCRIPTION:
The specific aims are (1) to test the feasibility and costs of methods and procedures for later use of MB-based combination therapy on a large scale, (2) to assess the safety of MB-based combination therapy, (3) to estimate the efficacy of MB-based combination therapy against malaria relapse, (4) to study the community acceptance of MB-based combination therapy, and (5) to strengthen the local capacity for malaria research and control in Jimma/Ethiopia.

Study design:

The study is designed as a pilot trial in adult patients with uncomplicated P. vivax malaria in Jimma, Ethiopia. Patients will be randomised to three treatment groups:

1. Arthemeter/Lumefantrine (AL)
2. AL-PQ, and
3. AL-MB. Follow-up will be over a period of 6 months.

Study population:

Adult patients with uncomplicated P. vivax malaria (age ≥18 years) in Jimma/Ethiopia (G6PD deficient subjects are excluded) will become enrolled in the outpatient departments of the study centres. The sample size will be 33 per study arm, a total of 99 patients.

Study treatments:

* AL standard treatments twice daily (total of 80 mg/dose A plus 480 mg/dose L) over first three study days
* PQ 15 mg once daily for 14 days
* MB 780 mg once daily for 14 days Treatments will be 100% directly observed.

Study outcomes:

Outcome parameters will be on feasibility and costs (e.g. recruitment rates, retention rates, costs per patient), on safety parameters (e.g. haemoglobin development during follow-up, incidence of adverse events), on efficacy parameters (e.g. incidence of P. vivax relapse during follow-up, malaria recurrence-free efficacy until day 180), and on community acceptance (e.g. perceptions on blue urine) during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Uncomplicated P. vivax monoinfection (asexual parasite count >250/µl)
* Axillary temperature ≥ 37.5°C or history of fever during last 48 hours
* Ability to tolerate oral drug therapy
* Written informed consent of patient
* Permanent residence in the study area

Exclusion Criteria:

* Therapy with an antimalarial (e.g. CQ, amodiaquine, pyrimethamine-sulfadoxine, quinine, any ACT) or an antibiotic which is effective against malaria parasites (e.g. doxycyclin, clindamycin, CoTrim) during last three weeks
* Mixed malaria infection
* Clinical danger signals (e.g. unable to stand or to sit, unable to drink, repeated vomiting, convulsions) or signs and symptoms of severe malaria (according to WHO definition)
* Known other serious illnesses (e.g. cardiac, renal, hepatic, pulmonary disease, severe malnutrition, severe infectious diseases)
* G6PD deficiency (<60% activity, WHO classification 1-3)
* Patients with known allergy to one or more of the study drugs
* Hemoglobin value <7 g/dL
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Study feasibility | 180 days
  Patient recruitment rates

SECONDARY OUTCOMES:
Incidence of P. vivax | 180 days
  Passive and active surveillance
Adverse events (AE) during total follow-up period | 180 days
  Passive and active surveillance
Study costs | 180 days
  Costs per patient

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Müller, Prof. Dr., Principal Investigator — Heidelberg University

IPD SHARING:
Plan to Share IPD: Undecided